CLINICAL TRIAL: NCT01566903
Title: Morphological and Dynamic Non Contrast-enhanced MR Angiography in the Exploration of Neurovascular Diseases
Brief Title: Neurovascular Non Contrast-Enhanced MR Angiography at 3T
Acronym: NCE MRA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A01258-33; LOC/11-19 (Other: Rennes University Hospital)
Record Dates: First submitted 2012-03-23; First posted 2012-03-29 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Neurovascular Diseases
Keywords: arterial stenosis; arteriovenous malformations; Post-treatment follow-up
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- arteriovenous malformations
- Arterial stenosis
- Post-treatment follow-up: Patient with an arteriovenous malformation for which treatment by embolization or radiosurgery is indicated

SUMMARY:
MR angiography (MRA) has become essential in the treatment of neurovascular diseases, including ischemic stroke - the first cause of disability in occidental countries, vascular malformations such as aneurysms, arteriovenous fistulas and malformations, whose treatments are improving year after year.

MRA is an alternative to digital substracted angiography (DSA), circumventing th use of endovascular catheterism, irradiation and injection of iodinated contrast agent. Contrast-Enhanced MRA (CE-MRA) with gadolinium injection is currently the reference standard for vascular MR exploration but still presents many limitations inherent to the injection of contrast medium. Hence, the synchronization of the acquisition with bolus contrast injection limits the improvement of spatial and temporal resolutions and requires an accurate synchronization of the acquisition with the arrival of the bolus.

Moreover, the acquisition can be repeated as required as it does not require any contrast injection.

Besides, the increase in nephrogenic systematic fibrosis clinical cases, which would be secondary to gadolinium chelates injection, in patients with chronic renal insufficiency has restricted the use of CE-MRA. More than 500 cases were described to date in the world.

Its occurrence is currently estimated around 4 % for patients in terminal chronic renal insufficiency and its mortality around 30 %.

According to the recommendations of AFSSAPS from August, 2007, two gadolinium contrast agent (Gadodiamide-OMNISCAN *, General Electric HealthCare and Gadopentetate Dimeglumine-MAGNEVIST *, Bayer HealthCare) are contraindicated if the glomerular filtration rate is lower than 30 ml/mn.

Non-contrast enhanced MR angiography (NCE MRA) techniques have been proposed to provide complete and non-invasive investigation of the vasculature, thus offering patients with chronic renal insufficiency, as well as pregnant or nursing women a surrogate with no side effects.

Moreover, the use of high field (3T) MR imaging offers improved signal to noise ratio. Combined with the use of phased array coils and parallel imaging, new NCE MRA sequences can achieve juxta-millimeter isotropic spatial resolution and temporal resolution of about 50 ms close to those of cerebral DSA.

These sequences allow a joint hemodynamical and morphological assessment of lesions, both at the cervical and cerebral levels, whether at diagnosis or during patient follow-up

DETAILED DESCRIPTION:
The main objective is to evaluate the quality of the NCE images obtained in the exploration of neurovascular diseases, at the cervical and cerebral levels.

Secondary objectives are:

* to compare the NCE MRA sequences with the CE MRA sequences used in the clinical routine.
* to evaluate the anatomic and hemodynamic changes observable with sequences in the follow-up of patients, particularly those treated with partial embolization or radiosurgery.

By circumventing the limitation to short bolus duration synchronization, the new dynamic sequences have the potential to achieve higher temporal resolution without compromising spatial resolution. Arteries and arteriovenous shunts may be more precisely identified and, due to a better visibility of small vessels allow a more accurate dynamic analysis.

Finally, the sequence being derived from arterial spin labeling, and differing from time of flight or phase contrast sequences, should allow for an exploration less dependent on the vascular geometry with better anatomical analysis. For example, the tendency to overestimate arterial stenoses could be reduced.

The robustness of sequences allow the non-invasive monitoring of patients including it possible to monitor the hemodynamic changes after radiosurgery or embolization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years
* Any adult patient known or clinically suspect to present a neurovascular disease (arterial stenosis ou arteriovenous malformations), the assessment of which requires an MRA or patient having an arteriovenous malformation for which treatment by embolization or radiosurgery is indicated multidisciplinary meeting and followed in the ordinary course of this treatment
* Patient able of accepting protocol information
* Patient who received information about the protocol and had not expressed its opposition to participate

Exclusion Criteria:

* A contraindication to MRI, in particular pacemakers or implantable defibrillators, cochlear implants, neurosurgical clips, intra-orbital or brain metallic foreign bodies, endo prothesis since less than 4 weeks or osteosynthesis material since less than 6 weeks
* Contraindication to the injection of contrast agent: pregnancy, lactation, history of allergic reaction to contrast agent injection
* Hemodynamically unstability, acute respiratory failure, a precarious condition or a need for continuous monitoring incompatible with the constraints of MR imaging
* Patient with severe kidney with Glomerular Filtration rate < 30 ml/min
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurovascular diseases
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-06-05 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
A reading grid assessing the image quality | 54 months
  Qualitative and quantitative evaluation of image quality :
  This analysis will be performed using a reading grid assessing the image quality (signal to noise ratio, motion artefacts, artefacts other than motion) and identifying the vessels visualized

SECONDARY OUTCOMES:
An evaluation grid classifying the main pathological findings | 54 months
  Assessment of diagnosis performance of the nem NCE MRA sequences :
  This assessment will be performed using an evaluation grid classifying the main pathological findings, ie arterial stenosis or arteriovenous shunts and assessing their extent
An evaluation of the performance of new sequences | 54 months
  Evaluation of the performance of new sequences to quantify hemodynamic parameters in arteriovenous shunts and detect anatomical and hemodynamic changes after treatment with partial embolization or radiosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: jean-yves gauvrit, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France